CLINICAL TRIAL: NCT00936403
Title: A Randomised, Open-labelled, Single Dose, Dose-escalation Trial Investigating Safety, Tolerability, Pharmacokinetics and Pharmacodynamics of Pegylated Long-acting Human Growth Hormone (NNC126-0083) Compared to Norditropin NordiFlex® in Growth Hormone Deficient Children
Brief Title: A Single Dose Trial in Growth Hormone Deficient Children Investigating Safety, Pharmacokinetics and Pharmacodynamics of Long Acting Growth Hormone
Status: Completed | Phase: Phase 2 | Type: Interventional
Sponsor: Novo Nordisk A/S (Industry)
Responsible Party: Sponsor
Allocation: Randomized | Model: Single Group | Masking: None | Purpose: Treatment
Other Study IDs: NN8630-1824; 2008-008240-25 (EudraCT Number)
Record Dates: First submitted 2009-07-09; First posted 2009-07-10 (Estimated); Last update posted 2017-02-08 (Estimated); Status verified 2017-02

CONDITIONS: Growth Hormone Disorder; Growth Hormone Deficiency in Children
MeSH Terms: interventions — NNC126-0083; Human Growth Hormone

STUDY DESIGN:
Oversight: Data Monitoring Committee: No

ARMS (2):
- NNC126-0083 (Experimental)
  Interventions: Drug: NNC126-0083
- Norditropin NordiFlex® (Active Comparator)
  Interventions: Drug: somatropin

INTERVENTIONS:
Drug: NNC126-0083 — One single dose administered in four dose levels in an escalating order
  Arms: NNC126-0083
Drug: somatropin — A daily dose of Norditropin NordiFlex® for seven days. Dose will remain constant
  Arms: Norditropin NordiFlex®

SUMMARY:
This trial is conducted in Europe. The aim of this clinical trial is to investigate the safety, tolerability, pharmacokinetics (the determination of the concentration of the administered medication in blood over time) and pharmacodynamics (the determination of the effect over time and the duration of action) of a long-acting growth hormone (NNC126-0083) in growth hormone deficient children.

ELIGIBILITY:
Inclusion Criteria:

* Confirmed diagnosis of growth hormone insufficiency as defined by two different GH provocation tests, defined as a peak of GH level less than 7ng/ml
* Pre-pubertal children
* Growth hormone replacement treatment for at least three months

Exclusion Criteria:

* Evidence of tumour growth or malignant disease
* Growth hormone deficient children with overt diabetes mellitus (fasting blood glucose more than 126mg/dl)

Ages: 6 Years to 12 Years | Sex: All | Healthy Volunteers: No
Age Groups: Child
Enrollment: 31 (Actual)
Dates: Start 2009-08; Primary Completion 2010-07 (Actual); Study Completion 2010-07 (Actual)

PRIMARY OUTCOMES:
Frequency of Adverse events (AEs) | 0-10 days after dosing

SECONDARY OUTCOMES:
AUC (0-168h), the area under the plasma NNC126-0083 profile in the interval 0-168 hours after trial product administration | Measured 10 days after dosing
IGF-I AUC (0-168h) the area under IGF-I profile in the interval 0-168 hours after trial product administration | Measured 10 days after dosing

CONTACTS AND LOCATIONS:
Overall Officials: Global Clinical Registry (GCR, 1452), Study Director — Novo Nordisk A/S
Locations (20):
- Belgium (2):
  - Novo Nordisk Investigational Site, Brussels
  - Novo Nordisk Investigational Site, Ghent
- Novo Nordisk Investigational Site, Prague, Czechia
- Novo Nordisk Investigational Site, Århus C, Denmark
- France (2):
  - Novo Nordisk Investigational Site, Bron
  - Novo Nordisk Investigational Site, Toulouse
- Israel (4):
  - Novo Nordisk Investigational Site, Beersheba
  - Novo Nordisk Investigational Site, Jerusalem
  - Novo Nordisk Investigational Site, Kfar Saba
  - Novo Nordisk Investigational Site, Petah Tikva
- Novo Nordisk Investigational Site, Skopje, North Macedonia
- Novo Nordisk Investigational Site, Ljubljana, Slovenia
- Spain (4):
  - Novo Nordisk Investigational Site, Barcelona
  - Novo Nordisk Investigational Site, Esplugues Llobregat
  - Novo Nordisk Investigational Site, Santiago de Compostela
  - Novo Nordisk Investigational Site, Vitoria-Gasteiz
- Turkey (Türkiye) (2):
  - Novo Nordisk Investigational Site, Ankara
  - Novo Nordisk Investigational Site, Istanbul
- United Kingdom (2):
  - Novo Nordisk Investigational Site, Birmingham
  - Novo Nordisk Investigational Site, Cambridge

REFERENCES:
- [Result] de Schepper J, Rasmussen MH, Gucev Z, Eliakim A, Battelino T. Long-acting pegylated human GH in children with GH deficiency: a single-dose, dose-escalation trial investigating safety, tolerability, pharmacokinetics and pharmacodynamics. Eur J Endocrinol. 2011 Sep;165(3):401-9. doi: 10.1530/EJE-11-0536. Epub 2011 Jul 1. PMID 21724838
- [Derived] Papathanasiou T, Agerso H, Damholt BB, Hojby Rasmussen M, Kildemoes RJ. Population Pharmacokinetics and Pharmacodynamics of Once-Daily Growth Hormone Norditropin(R) in Children and Adults. Clin Pharmacokinet. 2021 Sep;60(9):1217-1226. doi: 10.1007/s40262-021-01011-3. Epub 2021 Apr 17. PMID 33864240
- See also: Clinical Trials at Novo Nordisk — http://novonordisk-trials.com